CLINICAL TRIAL: NCT06895746
Title: Multi-omics Study in Citrin Deficiency for Characterization of Disease-specific Metabolites and Biomarker Identification
Brief Title: Multi-omics Study in Citrin Deficiency
Status: Active, not recruiting | Type: Observational
Sponsor: Johannes Haeberle (Other)
Collaborators: Citrin Foundation (Unknown); Bristol Royal Hospital for Children (Other); Central Manchester University Hospital NHS Foundation Trust (Unknown); University Hospital Birmingham NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); Mount Sinai Hospital, New York (Other); National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Pusan National University Yangsan Hospital (Other); Saitama Medical University (Other); Osaka Metropolitan University (Other); Tohoku University (Other); Kurume University (Other); University College London Hospitals (Other); Sheffield Children's NHS Foundation Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Kumamoto University (Other); Saiseikai Yokohama City Eastern Hospital (Other); Jikei University School of Medicine (Other); Yamagata University (Other); Chiba Children's Hospital (Unknown); Shinshu University Hospital (Unknown); Birmingham Women's and Children's NHS Foundation Trust (Other); National Hospital Organisation Hokkaido Medical Center (Unknown)
Responsible Party: Sponsor-Investigator, Johannes Haeberle, Head of Metabolic Laboratory, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: 2022-02306
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Citrin Deficiency
Keywords: citrin deficiency; multi-omics; biomarker identification
MeSH Terms: conditions — Adult-onset citrullinemia type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD patient: patients with citrin deficiency (mutation in SLC25A13 gene)
- healthy control: matched controls

SUMMARY:
Citrin deficiency (CD) is an underdiagnosed and understudied condition characterized by several distinct phenotypes: 1) neonatal intrahepatic cholestasis caused by citrin deficiency (NICCD), 2) the adaptation or silent period, 3) "failure to thrive and dyslipidemia" form of CD (FTTDCD), and 4) citrullinemia type II (CTLN2), with the latter representing the final and most severe form of the condition. There is currently no cure for CD and patients manage their symptoms with lifelong dietary intervention and regular checkups with their physicians. A major hurdle in developing effective treatments for CD is the lack of effective biomarkers that track well with disease severity or measure the effectiveness of therapeutics. The present study aims to identify robust circulating biomarkers of CD through analysis of blood samples from CD patients.

DETAILED DESCRIPTION:
Citrin deficiency (CD) is an inherited autosomal recessive metabolic condition that is also a secondary urea cycle disorder caused by mutations in the SLC25A13 gene, which encodes for the mitochondrial transporter, citrin. Citrin is a key component of the mitochondrial malate-aspartate shuttle (MAS) and is responsible for moving Nicotinamide Adenine Dinucleotide (NADH) from the cytosol into the mitochondria via reducing equivalents such as malate, which drives mitochondrial respiration to produce energy in the form of adenosine triphosphate (ATP). The MAS is also critical in regulating Nicotinamide Adenine Dinucleotide (NAD+/NADH) redox balance to maintain cytosolic redox-dependent metabolic pathways such as glycolysis, gluconeogenesis, amino acid metabolism, and lipid metabolism. Citrin is also required to supply cytosolic aspartate, which is the substrate of one of the urea cycle enzymes, namely argininosuccinate synthetase 1, and thus important for the proper functioning of the urea cycle.

The clinical presentations of citrin deficiency often vary widely between patients but can generally be distinguished by distinct clinical phenotypes, which are neonatal intrahepatic cholestasis caused by citrin deficiency (NICCD) that affects infants, the "failure to thrive and dyslipidemia" form of CD (FTTDCD) in childhood, the adaptation or silent period, and citrullinemia type II (CTLN2), which represents the most severe form of the condition. While only a small percentage of CD patients develop CTLN2, the prognosis for these patients is typically poor. It is notable that all CD patients above 1 year old (post-NICCD) naturally develop a characteristic food preference that favors a diet rich in protein and fat while being low in carbohydrates. Other clinical findings observed in some CD patients include fatty liver, fatigue, hypoglycemia, and failure to thrive.

There is currently no effective cure for CD. Before the onset of CTLN2, patients are primarily managed by diet control with a low carbohydrate, high protein and high-fat diet, as well as medium chain triglyceride (MCT) supplementation. CTLN2 patients have been treated with sodium pyruvate, arginine, and MCT with limited success, with severe cases requiring liver transplantation as the only solution. There are currently no specific biomarkers that effectively track the disease progression, making it challenging to monitor how well patients are actually doing or to measure the effectiveness of therapies. Without proper management or timely medical interventions, patients may develop CTLN2.

Given the urgent and unmet need for biomarkers specific to CD, the main goal of this study is to uncover disease-specific biomarkers by analyzing blood samples collected from CD patients using both targeted and untargeted metabolomics, proteomics, lipidomics, and transcriptomics. Targeted omics will involve the analysis of cellular pathways associated with the condition, such as the MAS pathway, glycolysis, protein metabolism, de novo lipogenesis, lipolysis, gluconeogenesis, NAD+ metabolism, ureagenesis, and the glutamine synthetase pathway. Identification of such biomarkers will allow a deeper understanding of the disease pathogenesis. Importantly, these biomarkers may enable better tracking of disease progression and may help to prevent the onset of CTLN2. Finally, these biomarkers will also greatly benefit the development of effective therapeutic options for CD in clinical trials by serving as measurable endpoints.

Obtaining the necessary material from patients consists of a minimally invasive venous blood sampling taken during a regular outpatient visit and after the informed consent of the patients or caretakers.

ELIGIBILITY:
Inclusion Criteria for patient group:

* confirmed diagnosis of citrin deficiency

Exclusion Criteria for control group:

* any metabolic disease

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Citrin deficiency (CD) is an inherited autosomal recessive metabolic condition that is also a secondary urea cycle disorder caused by mutations in the SLC25A13 gene, which encodes for the mitochondrial transporter, citrin.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
identification of biomarkers | three to five years from enrollment
  The primary endpoint is the identification of biomarkers from CD patient-derived blood samples that are expressed at levels significantly different from matched controls.

SECONDARY OUTCOMES:
biochemical profiles | three to five years from recruitment
  The secondary endpoint consists in the identification of unique biochemical profiles from CD patient-derived blood samples that are significantly different from matched controls, and the correlation with clinical condition and dietary regimen.

CONTACTS AND LOCATIONS:
Locations (23):
- Mount Sinai Hospital, New York, New York, United States
- Japan (11):
  - Kurume University, Kurume-shi, Fukuoka
  - Saitama Medical University, Saitama, Iruma
  - Saiseikai Yokohama City Eastern Hospital, Yokohama, Kanagawa
  - Jikei University Hospital, Tokyo, Minato City
  - Tohoku University, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - National Hospital Organisation Hokkaido Medical Center, Hokkaido, Sapporo
  - Osaka Metropolitan University, Osaka, Umeda
  - Chiba Children's Hospital, Chiba
  - Kumamoto University Hospital, Kumamoto
  - Yamagata University School of Medicine, Yamagata
- Pusan National University Yangsan Hospital, Yangsang, Gyeongsang, South Korea
- Taiwan (2):
  - Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (8):
  - Central Manchester University Hospital NHS Foundation Trust, Manchester, Lancashire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Birmingham Women's and Children's Hospital NHF Foundation Trust, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - University College London Hospital, London
  - Great Ormond Street Hospital for Children NHS foundation trust, London
  - Salford Royal NHS Foundation Trust, Salford
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes